CLINICAL TRIAL: NCT02993263
Title: Detection and Prediction of Postoperative Acute Myocardial Ischemic Injury/Infarction by the VectraplexECG System With CEB®
Brief Title: Postoperative Acute Myocardial Ischemic Injury
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was withdrawn as there was an ECG equipment and software malfunction. There is no results for this study because of the equipment malfunction.
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-1556
Record Dates: First submitted 2016-07-18; First posted 2016-12-15 (Estimated); Results first posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Noncardiac surgery (Other): VectraplexECG System with CEB® will be recorded after surgery and on day 1, 2 and 3 post operatively
  Interventions: Device: VectraplexECG System with CEB®

INTERVENTIONS:
Device: VectraplexECG System with CEB® — The device will be used after noncardiac surgery

SUMMARY:
The investigators propose to estimate the sensitivity and specificity of the VectraplexECG System for detecting acute myocardial ischemic injury, including acute myocardial infarctions after major non-cardiac surgery.

A 10 second CEB dynamic sequence recording will be obtained immediately after surgery in the post-anesthesia care unit.

On the first, second and third post operative morning a 10 second CEB dynamic sequence will be recorded. Blood will be sampled for troponin as well.

On the first, second and third post operative afternoons a 10 second CEB dynamic sequence will be recorded.

The morning 10 second CEB dynamic sequence and blood draw for troponin will continue as long as the patient remains hospitalized. The afternoon 10 second CEB dynamic sequence will continue as long as the patient remains hospitalized.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. ≥ 45 years old.
3. Anticipated hospitalization of at least two nights.

Exclusion Criteria:

1. Inadequate ECGs, based on an initial 10-second trace, as defined by:

   * wandering baseline
   * excessive noise
   * ventricular ectopy
   * pacer spikes or
   * lead placement error
2. Atrial fibrillation.
3. Average heart rate exceeding 90 beats/minute.
4. Evidence of previous myocardial infarction:

   * Pathologic Q waves (≥0.04 sec) and/or
   * Pathologic findings of a healed or healing MI and/or
   * Evidence from an imaging study of a region of loss of viable myocardium

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-05-14 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Sessler, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment process started by screening patients who are scheduled for non cardiac surgery. These patients are approached during their anesthesia clearance visit.
Pre-assignment Details: Open label study
Groups:
- Noncardiac Surgery: VectraplexECG System with CEB® used after surgery and on day 1, 2, and 3 postoperatively
Period: Overall Study
Arm/Group | Noncardiac Surgery
Started | 323
Completed | 0
Not Completed | 323
Not completed — Equipment Software failed and results were lost. | 323

BASELINE CHARACTERISTICS:
Arm/Group | Noncardiac Surgery
Number analyzed (Participants) | 323
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 164
  Male | 159
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Accuracy
Description: Accuracy of VectraplexECG System with CEB
Time Frame: 1 minute to complete the test
Population: Data were not collected, because of the malfunction of the equipment software failed.
Arm/Group | Noncardiac Surgery
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 30 days
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Noncardiac Surgery
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-01): https://cdn.clinicaltrials.gov/large-docs/63/NCT02993263/Prot_SAP_000.pdf